CLINICAL TRIAL: NCT07321431
Title: The Optimal Measurement Time for the New Gallbladder Function Assessment Method: A Prospective, Multicenter, Double-Blind, Crossover Trial
Brief Title: The Optimal Measurement Time for the New Gallbladder Function Assessment Method
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Director of Surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: GB evaluating
Record Dates: First submitted 2025-12-13; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Gallbladder; Functional Disturbance
Keywords: Gallbladder Contractile Function; Ultrasound Examination; Olive oil; Protein Bar; Optimal time
MeSH Terms: interventions — Olive Oil

STUDY DESIGN:
Intervention Model Description: A two-period crossover design will be adopted, in which the two intervention methods will be randomly assigned.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI, study biostatistician will be masked until database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fried eggs (Experimental): First, the intervention of oral administration of 2 fried eggs is carried out. The size of the gallbladder is evaluated by ultrasound examination. The washout period is 1 week. After that, the first intervention process of group B is repeated.
  Interventions: Dietary Supplement: oral administration of 2 fried eggs
- protein bars (Active Comparator): First, an intervention with oral protein bars + 50ml olive oil is conducted. The size of the gallbladder is evaluated through ultrasound examination. The washout period is 1 week. After that, the first intervention process of Group A is repeated.
  Interventions: Dietary Supplement: oral protein bars + 50ml olive oil

INTERVENTIONS:
Dietary Supplement: oral administration of 2 fried eggs — First, the intervention of oral administration of 2 fried eggs is carried out. The size of the gallbladder is evaluated by ultrasound examination. The washout period is 1 week. After that, the first intervention process of group B is repeated.
  Arms: fried eggs
Dietary Supplement: oral protein bars + 50ml olive oil — First, an intervention with oral protein bars + 50ml olive oil is conducted. The size of the gallbladder is evaluated through ultrasound examination. The washout period is 1 week. After that, the first intervention process of Group A is repeated.
  Arms: protein bars

SUMMARY:
This is a multicenter, prospective, randomized, double-blind, crossover study involving healthy individuals, aiming to evaluate the stability of oral protein bars + olive oil as a new method for determining gallbladder contraction function and its optimal diagnostic time window.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, single-blind, crossover study involving healthy individuals. This study will use a crossover trial method to compare oral fried eggs with oral protein bars + olive oil. Gallbladder ultrasound examinations will be performed at different time points to measure gallbladder volume, and the changes in gallbladder contraction rates at different time points under the two interventions will be calculated to determine the optimal time window for assessing gallbladder contraction function. On the other hand, the investigators will verify the stability of oral protein bars plus olive oil as a new method for measuring gallbladder contraction function, evaluate its reliability and reproducibility across different regions, hospitals, and populations, ensure its wide clinical application, and provide stronger support for the diagnosis and treatment of gallbladder-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound assessment identifies people with normal biliary tract structure.

Exclusion Criteria:

* History of Endoscopic Retrograde Cholangiopancreatography
* Previous gallstone removal surgery with gallbladder preservation
* Other biliary tract diseases and related surgical history
* History of acute or chronic pancreatitis
* History of gastrointestinal surgery
* Gastrointestinal obstruction
* Dysfunction of the sphincter of Oddi
* Gallbladder neck polyps
* Abnormal gallbladder structure
* Gallbladder mass
* Biliary infection or stones
* Congenital biliary abnormalities
* Biliary injury or surgery
* Biliary tumors
* Gastrointestinal bleeding, liver cirrhosis, or other malignant diseases
* Significant arrhythmia, bradycardia, or atrioventricular block
* Severe hypertension, liver or kidney insufficiency
* Immune, endocrine, hematological, or mental disorders
* Severe cerebrovascular disease
* Allergy to relevant foods
* Pregnant or breastfeeding women
* Unwillingness or inability to consent to participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Gallbladder Volume | during procedure
  Formula for Ultrasound Measurement of Gallbladder Volume (L × W × D × 0.52). Measurements were taken every 20 minutes starting from 30 minutes after the intervention, with a total of 5 measurements (i.e., the gallbladder volume was measured at 30 minutes, 50 minutes, 70 minutes, 90 minutes, and 110 minutes respectively).
Gallbladder contraction rate | during procedure
  Subtract the volume of the gallbladder after intervention from the volume of the gallbladder on an empty stomach, then divide by the volume of the gallbladder on an empty stomach, and finally multiply by A-B/A%. The gallbladder contraction rate was calculated at all the above time points.

SECONDARY OUTCOMES:
Presence of Abdominal | 30 days
  Pain Post-Intervention If abdominal pain is present, it will be assessed using the Numerical Rating Scale (NRS) within 0-10, The higher the score, the more serious it is.
Occurrence of Acute Pancreatitis | 30 days
  Post-Intervention Pain and Amy 3 times as normal.
Occurrence of Gastrointestinal Bleeding Post-Intervention | 30 days
  Black stool or decrease of hemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D. Ph. D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (5):
- China (5):
  - Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu
  - The First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Jinqiu Hospital of Liaoning Province, Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Honghui Hospital of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ai XN, Wang TF, Zhang Q, Ouyang CG, Wu ZY. Changes in Gallbladder Contractile Function and its Influencing Factors After Minimally Invasive Gallbladder-Preserving Surgery for Cholecystitis With Incarcerated Gallstones. Front Surg. 2022 Jul 14;9:926141. doi: 10.3389/fsurg.2022.926141. eCollection 2022. PMID 35910468
- [Background] Rehfeld JF. Clinical endocrinology and metabolism. Cholecystokinin. Best Pract Res Clin Endocrinol Metab. 2004 Dec;18(4):569-86. doi: 10.1016/j.beem.2004.07.002. PMID 15533776